CLINICAL TRIAL: NCT06321692
Title: Early Identification of Cardiac Involvement in Patients With Carcinoid: Clinical and Prognostic Implications
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IEO 1003
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation of blood levels of biomarkers of cardiac damage (Other): Evaluation of blood levels of biomarkers of cardiac damage (ultra-sensitive troponin I), hemodynamic impairment (BNP, NT-proBNP), and cardiac fibrosis (ST2) in patients with diagnosed neuroendocrine tumours (NET) with or without carcinoid syndrome
  Interventions: Other: Evaluation of blood levels of biomarkers of cardiac damage

INTERVENTIONS:
Other: Evaluation of blood levels of biomarkers of cardiac damage — Evaluation of ultra-sensitive troponin I, BNP, NT-proBNP, and ST2 in patients with diagnosed neuroendocrine tumours (NET) with or without carcinoid syndrome

SUMMARY:
This study is for patients with neuroendocrine tumours (NET) with or without carcinoid syndrome followed by NET Unit of European Institute of Oncology.

The objective of the trial is to evaluate biochemical markers of myocardial injury (high-sensitive troponins), haemodyinamic markers (pro-brain natriuretic peptide (BNP), N-terminal (NT)-BNP (NT-proBNP)), and markers of fibrosis (Suppression of Tumorigenicity 2 (ST2) in patients with neuroendocrine tumours (NET) with or without carcinoid syndrome.

DETAILED DESCRIPTION:
The main aim of this study is to evaluate blood levels of biomarkers of cardiac damage (ultra-sensitive troponin I), hemodynamic impairment (BNP, NT-proBNP), and cardiac fibrosis (ST2) in patients with diagnosed neuroendocrine tumours (NET) with or without carcinoid syndrome The secondary objective is to correlate the levels of the above markers with the presence/entity of cardiac involvement and its progression over time.

All patients will undergo:

* a baseline assessment including:

  * blood sampling for US-Troponin I, BNP, NT-proBNP, ST2
  * cardiological evaluation including ECG and echocardiogram
* a three-monthly revaluation of these markers
* a six monthly cardiological reassessment with a echocardiogram

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with metastatic NET with or without carcinoid referred to the Unit of Neuroendocrine Tumors of European Institute of Oncology

Exclusion Criteria:

* age <18 years
* patients diagnosed with heart disease prior to diagnosis of NET

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-10-09 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
blood levels of biomarkers of cardiac damage | 3 months
  Evaluation of blood levels of ultra-sensitive troponin I
blood levels of biomarkers of hemodynamic impairment | 3 months
  Evaluation of blood levels of BNP, NT-proBNP
blood levels of biomarkers of cardiac fibrosis | 3 months
  Evaluation of blood levels of ST2

SECONDARY OUTCOMES:
Correlation between the levels of the biomarkers and the presence/entity of cardiac involvement | 6 months
  Correlation between the levels of the biomarkers and echocardiographic features to define cardiac involvement.
  The features considered to define the cardiac involvement will beù
  * Tricuspid valve regurgitation, ranging from mild to severe
  * Pulmonary valve regurgitation and/or stenosis
  * Dilated right atrium
  * Dilated right ventricle
  * Reduced right ventricular function

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Cardinale, MD, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy